CLINICAL TRIAL: NCT00339911
Title: Collection and Distribution of Samples From Healthy Donors for In Vitro Research at NCI-Frederick
Brief Title: Collection and Distribution of Samples From Healthy Donors for In Vitro Research at the NCI-Frederick
Status: Enrolling by invitation | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999999046; OH99-C-N046
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2025-12-24 (Actual); Status verified 2025-07-09

CONDITIONS: Healthy Donors
Keywords: Repository; Phlebotomy; Venipuncture; Anemia; Occupational Health Services; Natural History
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1/ single cohort: Healthy NCI Frederick Cancer Research and Development Center employees

SUMMARY:
Background

-NCI-Frederick scientists performing in vitro studies involving human specimens have a need for a reliable and consistent source of samples which protects the donor from research risks.

Objective

-The purpose of this protocol is to establish a centralized repository for the collection and distribution of samples (either blood, buccal mucosal cells, semen, urine, or nail clippings) from paid, healthy volunteer donors for in vitro research conducted by NIH investigators located at NCI-Frederick and Ft. Detrick. Research will include, but are not limited to, genotype analysis, immune function studies, drug screening, vaccine development, method development, quality control testing of reagents, and propagation of infectious agents, including HIV.

Eligibility:

Healthy NCI-Frederick employees and other NIH staff located at Ft. Detrick will be recruited. Potential donors will be excluded if screening indicates exposure to HIV, HTLV, Hepatitis C or Hepatitis B virus infection.

Study Design:

Investigators requesting to participate to the Research Donor Program (RDP) by receiving samples for research use will be required to submit a written memo of request, briefly describing the nature of the research and providing assurance that samples provided through this protocol will be used solely for in vitro research.

These Investigators will receive samples that will be either anonymous or coded, depending on the specific need.

Codes will be securely maintained and under no circumstances will donor identity be released to Investigators.

Donors will receive financial compensation for their time, discomfort and inconvenience according to an established schedule; compensation for blood donation is based on the volume donated.

DETAILED DESCRIPTION:
Background

-NCI-Frederick scientists performing in vitro studies involving human specimens have a need for a reliable and consistent source of samples which protects the donor from research risks.

Objective

-The purpose of this protocol is to establish a centralized repository for the collection and distribution of samples (either blood, buccal mucosal cells, semen, urine, feces, nasopharyngeal swabs, or nail clippings) from paid, healthy volunteer donors for in vitro research conducted by NIH investigators located at NCI-Frederick and Ft. Detrick. Research will include, but are not limited to, genotype analysis, immune function studies, drug screening, vaccine development, method development, quality control testing of reagents, and propagation of infectious agents, including HIV.

Eligibility:

Healthy NCI-Frederick employees and other NIH staff located at Ft. Detrick will be recruited. Potential donors will be excluded if screening indicates exposure to HIV, HTLV, Hepatitis C or Hepatitis B virus infection.

Study Design:

Investigators requesting to participate to the Research Donor Program (RDP) by receiving samples for research use will be required to submit a written memo of request, briefly describing the nature of the research and providing assurance that samples provided through this protocol will be used solely for in vitro research.

These Investigators will receive samples that will be either anonymous or coded, depending on the specific need.

Codes will be securely maintained and under no circumstances will donor identity be released to Investigators.

Donors will receive financial compensation for their time, discomfort and inconvenience according to an established schedule; compensation for blood donation is based on the volume donated.

ELIGIBILITY:
* INCLUSION CRITERIA:

Individuals must meet the following eligibility criteria to be entered into the RDP donor pool, as follows:

1. Age 18 or older.
2. Weight of 110 lb or greater.
3. All subjects must have the ability and agree to participate fully and comply with the procedures of the protocol and provide informed consent.
4. Registration for participation in semen donation is limited to males currently enrolled in the donor pool.
5. Subjects must be NCI Frederick Employees

EXCLUSION CRITERIA:

Individuals with any of the following will be excluded from the donor pool:

1. History of chronic illness that might increase the risks associated with phlebotomy, including but not limited to heart, lung, or kidney disease
2. Current acute illness.
3. History of clotting disorders.
4. Current medications which might increase the risk associated with phlebotomy.
5. History of syncope or other difficulty with venipuncture.
6. Anemia, as determined by hematocrit or hemoglobin.

   Hematocrit acceptable range for males: 40-51 percent.

   Hematocrit acceptable range for females: 34-46 percent.
7. Hemoglobin acceptable range for males: 12.5-17.0 g/dl

   Hemoglobin acceptable range for females: 11.5-15.2 g/dl
8. Positive blood test for exposure to HIV-1, HIV-2, HTLV-1, HTLV-2, or HCV or for HBV surface antigens.
9. Individuals whose activities or conditions place them at high risk of HIV infection are asked not to donate.
10. Males who qualify for participation in the donor pool will be excluded from participation in semen donation if they have knowingly had any injury, infection, or treatment performed that renders them incapable of producing sperm.
11. Pregnancy: Pregnant women will not be allowed to enroll in this study because there is no benefit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy NCI Frederick Cancer Research and Development Center employees@@@@@@
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 1999-11-01 (Actual); Primary Completion 2030-10-01 (Estimated); Study Completion 2030-10-13 (Estimated)

PRIMARY OUTCOMES:
Establish a centralized repository for the collection and distribution ofsamples | Ongoing
  Collection of biospecimens

CONTACTS AND LOCATIONS:
Overall Officials: Janelle Cortner, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- NCI Frederick Cancer Research Center, Frederick, Maryland, United States

REFERENCES:
- [Background] Merz JF, Sankar P, Taube SE, Livolsi V. Use of human tissues in research: clarifying clinician and researcher roles and information flows. J Investig Med. 1997 Jun;45(5):252-7. No abstract available. PMID 9249997
- [Background] McLeod BC, Price TH, Owen H, Ciavarella D, Sniecinski I, Randels MJ, Smith JW. Frequency of immediate adverse effects associated with apheresis donation. Transfusion. 1998 Oct;38(10):938-43. doi: 10.1046/j.1537-2995.1998.381098440858.x. PMID 9767744